CLINICAL TRIAL: NCT07221812
Title: Continuous Glucose Monitors (CGMs) and Readmission Rates
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HP-00116128
Record Dates: First submitted 2025-10-06; First posted 2025-10-28 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Diabetes (DM)
Keywords: Continuous Glucose Monitors
MeSH Terms: conditions — Diabetes Mellitus | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Real time-CGM (Experimental): The Real Time-CGM Group will wear the Dexcom G7 CGM device. Their glucose data will be shared in real-time to health care providers for subsequent treatment decisions.
  Interventions: Device: Continuous Glucose Monitor
- Point of Care (POC) (Other): The Point of Care (POC) group will use "finger sticks" to assess blood glucose values.
  Interventions: Other: Control Group

INTERVENTIONS:
Device: Continuous Glucose Monitor — The Dexcom G7 (real-time data) will be placed on all individuals randomized to the Intervention group. Their data will be shared with health care providers using a CGM software application. Providers will use this information during scheduled contact visits to make treatment decisions.
  Arms: Real time-CGM
Other: Control Group — The control group will use "finger sticks", usual Point of Care (POC), to measure blood glucose values. This information will be shared with providers and used for all treatment decisions at scheduled visits.
  Arms: Point of Care (POC)

SUMMARY:
Among the diffident groups of patients, those with chronic and severe medical conditions are more likely to be readmitted to the hospital. It is not surprising therefore that patients with diabetes have high readmission rates. Patients with diabetes have 40% higher re-hospitalization rates compared with those patients without diabetes, with 30-day readmission rates reported to range between 14% and 26%. It should be noted that almost 30% of the patients with diabetes are experiencing two or more hospital admissions per year, accounting for more than 50% of total hospitalizations and hospital health care costs. This research application will evaluate whether the initiation of Continuous Glucose Monitor (CGM) devices at the time of hospital discharge will lead to better glucose control and health outcomes compared to the use of "finger sticks" Point of Care (POC) following hospital discharge among patients with diabetes. This study will be a two arm (Real Time CGM vs POC) single center RCT at the Baltimore VA Medical Center. One hundred and twenty individuals will be recruited and randomly assigned (1:1) to either Real Time CGM or to POC following hospital discharge. All subjects will be followed from for 3 months post hospital discharge.

DETAILED DESCRIPTION:
Utilizing CGM devices for patients with diabetes at hospital discharge can be a feasible and easily to implement intervention, improving glycemic control. Compared to Point of Care (POC) glucose testing, CGM devices can provide an easier and painless method for monitoring blood glucose levels. By checking glucose values every couple of minutes, having alarm features and by having the ability to provide remote glucose monitoring (with software applications -smartphones-Bluetooth and internet), CGMs can have many benefits for patients with diabetes following hospital discharge: They can help patients with diabetes and their providers to achieve better glucose control after hospital discharge, reducing hyperglycemia, hypoglycemia and glucose variability, conditions that are associated with adverse outcomes among patients with diabetes. As extreme glucose values (hyperglycemia -hypoglycemia- glucose variability) are more common during illness in patients with diabetes, frequent glucose monitoring by CGMs can help patients as also medical providers to utilize them as another "vital sign", leading to early interventions.

These early interventions can have many other potential beneficial health effects. By monitoring glucose values closely, they can decrease hyperglycemia and hypoglycemia leading to better glucose control, reduced post discharge complications and as a result decrease readmission rates and mortality. Hospital readmissions, especially when they occur during the early period after hospital discharge, represent a marker of poor-quality healthcare delivery and have been associated with increased health care costs. In an effort to reduce readmission rates, the Centers for Medicare and Medicaid Services (CMS) Readmissions Reduction Program penalizes hospitals with high 30-day readmission rates. Among patients, those with diabetes have high readmission rates, ranging between 14% and 26%. This is translated to increased hospital expenses: It has been estimated that the cost of 30-day readmissions for patients with diabetes is nearly $25 billion. In addition, using CGM devices early upon discharge can lead to decreasing Emergency Department (ED) visits and post discharge mortality.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age
2. Patients with diabetes who are anticipated to be treated with any type of insulin after hospital discharge and with or without non-insulin medications (excluding those who are expected to be treated with correctional-sliding scale insulin regimens only
3. Uncontrolled glycemic control, defined as hyperglycemia with HbA1c ≥8%

Exclusion Criteria:

1. Patients with diabetes who are anticipated to be treated with diet only, any combination of non-insulin antidiabetic drugs only, sliding scale correctional insulins (with or without non-insulin medications) after hospital discharge.
2. Patients at the time of screening on insulin pumps or CGMs
3. Pregnant patients
4. Patients with extensive skin disease or allergies that preclude wearing the CGM sensor
5. Patients without current access of (or who are unable to obtain) a smartphone device and internet
6. Patients who have end-stage renal disease requiring dialysis
7. Patients with significant psychiatric illness or any other condition which by investigator decision makes the subject incapable of understanding the objectives and potential consequences of the study
8. taking hydroxyurea
9. Employed by, or having immediate family members employed by Dexcom, or having a direct supervisor at place of employment who is also directly involved in conducting the clinical trial (as a study investigator, coordinator, etc.); or having a first-degree relative who is directly involved in conducting the clinical trial

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-11-18 (Estimated); Primary Completion 2027-11-17 (Estimated); Study Completion 2028-11-17 (Estimated)

PRIMARY OUTCOMES:
Change in glycemic control | 90 days
  HbA1c
Change in hypoglycemia events | 90 days
  Hypoglycemia < 70 mg/dL
Change in Glucose Variability | 90 days
  Glucose Variability- Coefficient of Variation (CV%)
Change in Time In Range (TIR) | 90 days
  Change TIR (70-180 mg/dL)
Change in Glycemic Risk Index (GRI) | 90 days
  GRI (Hyperglycemia Component/Hypoglycemia Component)
Change in average glucose values at 90 days post discharge. | 90 days
  Change in Average glucose values (mg/dL)

SECONDARY OUTCOMES:
Change in 30-day readmission rates | 30 days
  Change in readmission rates
Change in 60-day readmission rates | 60 days
  Change in 60-day admission rates
Change in 90-day readmission rates | 90 days
  Change in 90-day readmission
Change in Emergency Department (ED) visits at 30-days | 30 days
  Change in ED visits at 30 days
Change in ED visits at 60 days | 60 days
  Change in ED visits at 60 days
Change in ED visits at 90 days | 90 days
  Change in ED visits at 90 days
Change in Mortality rates at 30 days | 30 days
  Change in Mortality rates at 30 days
Change in mortality rates at 60 days | 60 days
  Change in mortality rates at 60 days.
Change in mortality rates at 90 days | 90 days
  Change in mortality rates at 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Ilias Spanakis, MD, Principal Investigator — Baltimore VA Medical Center
Locations (1):
- Baltimore VA Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
IPD information is not necessary to share our study findings to the sponsor or peer-review organizations